CLINICAL TRIAL: NCT02369744
Title: Comparison of Silodosin vs. Tamsulosin on Spontaneous Passage of Acutely Obstructing Ureteral Calculi in Medical Expulsive Therapy
Brief Title: Silodosin Versus Tamsulosin for Treatment of Ureteral Stones
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: due to lack of suitable patient population
Sponsor: Albert Einstein Healthcare Network (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HN 4441
Record Dates: First submitted 2014-06-19; First posted 2015-02-24 (Estimated); Results first posted 2020-03-19 (Actual); Last update posted 2020-06-23 (Actual); Status verified 2017-05

CONDITIONS: Ureteral Calculus; Ureterolithiasis; Ureteral Stone
Keywords: Ureteral calculus; Ureterolithiasis; Ureteral stone; Kidney stone; Medical expulsive therapy; tamsulosin; silodosin; rapaflo; flomax
MeSH Terms: conditions — Ureteral Calculi; Ureterolithiasis; Kidney Calculi | interventions — silodosin; Tamsulosin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Silodosin (Active Comparator): Subjects in the Silodosin Group will be given silodosin 8 mg tablets, one tablet to be taken PO each day for two weeks.
  Interventions: Drug: Silodosin
- Tamsulosin (Active Comparator): Subjects in the Tamsulosin Group will be given tamsulosin 0.4 mg tablets, one tablet to be taken PO each day for two weeks.
  Interventions: Drug: Tamsulosin

INTERVENTIONS:
Drug: Silodosin — 8mg tablet, 1 tab PO daily for 2 weeks
  Other Names: Rapaflo
  Arms: Silodosin
Drug: Tamsulosin — 0.4 mg Tab, 1 tab PO daily for 2 weeks
  Other Names: Flomax
  Arms: Tamsulosin

SUMMARY:
Ureteral calculi, commonly known as kidney stones, are a frequent cause of Emergency Department (ED) visits. These stones can get caught in the ureter (the tube connecting the kidney to the bladder) and cause symptoms including pain, nausea, and vomiting. As long as the obstructing stone meets certain conditions and the patient isn't too sick, the patient is usually sent home to try and pass the stone without surgery. This treatment is known as medical expulsive therapy (MET), and routinely involves the use of a drug called tamsulosin, which relaxes the smooth muscle of the urinary system to help the stone pass. Silodosin is a drug in the same class of tamsulosin, but which is thought to have a more selective action and a quicker onset, which would theoretically make it better for aiding in kidney stone passage. The purpose of this study is a head-to-head, blinded comparison of these two drugs to see how quickly they result in stone passage. Subjects are patients presenting to the ED with acute kidney stone shown by CT scan, and who are appropriate for MET. The main study intervention is randomization to receiving either tamsulosin or silodosin. The hypothesis is that silodosin will have decreased time to stone passage compared to tamsulosin.

Subjects who qualify and consent are randomized to a two-week course of either silodosin or tamsulosin. They are also given prescriptions for standard of care medications for pain and nausea, as well as a pain diary. They receive a follow-up phone call after one week to remind them of their follow-up appointment, ask about adverse events, and determine if their stone has passed. They have a follow-up visit with study staff at the end of their two week treatment to collect their pain diary, pill count, adverse events, and to determine if their stone has passed. Study participation ends after this follow-up visit.

DETAILED DESCRIPTION:
Procedures Involved in the Research. This study is a prospective, randomized, double-blinded, head-to-head trial comparing two medications. Patients with symptoms of renal colic who present to the emergency department will be evaluated by the ED staff as per usual routine. After a work-up (including routine chemistry, complete blood count, urine analysis, urine culture, and non-contrast CT scan of the abdomen and pelvis) has been completed, patients who meet inclusion criteria will be asked whether they are willing to enroll in the study. Those who are unsuitable for the study or unwilling to participate will continue to receive routine care for their ureteral calculus. Those who consent will be enrolled as subjects in the study, and given a 2-week supply of either tamsulosin or silodosin in blinded bottles with the appropriate dosing instructions. The prescriptions will be dispensed by the pharmacy; therefore the subjects and study staff will be blinded to which prescription the subject receives. Randomization will be done in advance and a key made to correlate subject enrollment number with which prescription they have received. Throughout the study, the study staff will make no efforts to ascertain which medication the subject has been given, unless an adverse event is suspected. Each participant will be given an information card that details the two possible medications they are taking, which can be presented to their physicians as needed.

Subjects will then be discharged to home as per routine care with instructions to drink plenty of fluids, and will be given a strainer and asked to attempt to catch their ureteral calculus. They will also be given a standardized prescription analgesic package (Percocet 5/325mg #20, Motrin 600mg #60, Zofran OD 4mg #20 with standard dosing instructions) and a Visual Analog Pain Scale diary to be filled out daily. Subjects will be given standardized discharge instructions as per standard of care that will include indications for immediate ED return for signs and symptoms of infection or MET failure (fever, worsening pain, vomiting, lethargy, unsteadiness, syncope or inability to tolerate oral pain medications). As per standard of care, they will be instructed to return to the ER immediately if they develop any of these symptoms. Finally, the subject's contact information will be collected at the time of enrollment and a follow-up appointment will be scheduled for them with Urology in 4 weeks to ensure they get appropriate and timely specialty follow-up. This follow-up is also standard of care, and will occur after the subject's participation in the study ends.

Each subject will be scheduled to return to the ER in 2 weeks to be seen by the research staff for data collection. They will be asked to bring their pill bottle and visual analog pain scale diary to this visit. If the subject reports having passed a stone consistent with their initial imaging, or have resolution of their pain to suggest they passed the stone unseen, this will conclude their participation in the study. However, if they are still having symptoms, their case will be categorized as an outpatient treatment failure and the subject will be registered to be seen by an ER Physician and a Urology consult will be ordered, concluding their participation in the study. This is current standard of care, and will be covered by insurance. Any subject that has an unscheduled visit to an ER for a ureterolithiasis-related complaint will also be considered an outpatient treatment failure. This will also conclude their participation in this study.

To ensure follow-up, subjects will be called one week after enrollment. They will be reminded of their 2-week follow-up appointment and the need to bring in their pill bottles. Each subject will also be asked if they have passed the stone or had resolution of the pain. The will be reminded that they must follow-up even if they are no longer having symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Adults age 18 to 70 years
* Non-diabetic
* Unilateral ureteral calculus 4 to 10 mm visible on CT scan within the ureter
* Serum creatinine level within normal range
* Ability to tolerate oral fluids and oral pain medication
* Ability to make informed medical decisions regarding consent
* Willingness to follow up in the ER in two weeks

Exclusion Criteria:

* Adults unable to consent
* Age <18
* Signs of infection including Temperature >38º C or Urinalysis with any of the following: Positive Leukocyte Esterase, Positive Nitrates, or White Blood Cell Count >5/hfp in the setting of a positive urine culture (defined as a single isolated bacterial species population of >100,000 CFU)
* Patients with chronic pain already undergoing treatment with narcotic medications
* Patients already taking an alpha adrenergic antagonist medication
* Pregnant women
* Prisoners
* No working phone number

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2013-03; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Boroughf, DO, Principal Investigator — Einstein Healthcare Network; James Gardner, MD, Principal Investigator — Einstein Healthcare Network
Locations (1):
- Einstein Medical Center Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hollingsworth JM, Rogers MA, Kaufman SR, Bradford TJ, Saint S, Wei JT, Hollenbeck BK. Medical therapy to facilitate urinary stone passage: a meta-analysis. Lancet. 2006 Sep 30;368(9542):1171-9. doi: 10.1016/S0140-6736(06)69474-9. PMID 17011944
- [Background] Parsons JK, Hergan LA, Sakamoto K, Lakin C. Efficacy of alpha-blockers for the treatment of ureteral stones. J Urol. 2007 Mar;177(3):983-7; discussion 987. doi: 10.1016/j.juro.2006.10.023. PMID 17296392
- [Background] Pedro RN, Hinck B, Hendlin K, Feia K, Canales BK, Monga M. Alfuzosin stone expulsion therapy for distal ureteral calculi: a double-blind, placebo controlled study. J Urol. 2008 Jun;179(6):2244-7; discussion 2247. doi: 10.1016/j.juro.2008.01.141. Epub 2008 Apr 18. PMID 18423747
- [Background] Steinberg PL. Re: Karim Bensalah, Margaret Pearle and Yair Lotan. Cost-effectiveness of medical expulsive therapy using alpha-blockers for the treatment of distal ureteral stones. Eur urol 2008;53:411-9. Eur Urol. 2008 Aug;54(2):469; author reply 469. doi: 10.1016/j.eururo.2008.01.077. Epub 2008 Feb 4. No abstract available. PMID 18281146
- [Background] Hermanns T, Sauermann P, Rufibach K, Frauenfelder T, Sulser T, Strebel RT. Is there a role for tamsulosin in the treatment of distal ureteral stones of 7 mm or less? Results of a randomised, double-blind, placebo-controlled trial. Eur Urol. 2009 Sep;56(3):407-12. doi: 10.1016/j.eururo.2009.03.076. Epub 2009 Apr 3. PMID 19375849
- [Background] Preminger GM, Tiselius HG, Assimos DG, Alken P, Buck AC, Gallucci M, Knoll T, Lingeman JE, Nakada SY, Pearle MS, Sarica K, Turk C, Wolf JS Jr; American Urological Association Education and Research, Inc; European Association of Urology. 2007 Guideline for the management of ureteral calculi. Eur Urol. 2007 Dec;52(6):1610-31. doi: 10.1016/j.eururo.2007.09.039. No abstract available. PMID 18074433
- [Background] Kobayashi S, Tomiyama Y, Hoyano Y, Yamazaki Y, Sasaki S, Kohri K. Effects of silodosin and naftopidil on the distal ureter and cardiovascular system in anesthetized dogs: comparison of potential medications for distal ureteral stone passage. J Urol. 2010 Jan;183(1):357-61. doi: 10.1016/j.juro.2009.08.106. PMID 19914658
- [Background] H Lepor et al. Double-Blind, Randomized, Parallel-Group Study To Define Electrocardiographic Effects Of Silodosin. Journal of Urology 179(4), May 2008

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 0 Participants analyzed. PI has left the institution. Efforts made to contact the PI were unsuccessful. No study data available
Pre-assignment Details: 0 Participants analyzed. PI has left the institution. Efforts made to contact the PI were unsuccessful. No study data available
Period: Overall Study
Arm/Group | Silodosin | Tamsulosin
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 0 Participants analyzed. PI has left the institution. Efforts made to contact the PI were unsuccessful. No study data available
Groups:
- Total: Total of all reporting groups
Arm/Group | Silodosin | Tamsulosin | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical
Age, Continuous
Sex: Female, Male
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Time to Stone Passage
Description: The primary outcome measure will be the time it takes for the stone to pass. Stone passage will be defined as the subject self-reporting passage of a stone that is consistent with their imaging, or resolution of their pain to suggest unseen passage of their stone. This outcome will be measured from the initial emergency department visit, and gathered at the one-week follow-up call as well as the two-week follow-up visit.
Time Frame: at 2 weeks
Population: Data is not available
Arm/Group | Silodosin | Tamsulosin
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Use of Pain Medication
Description: The subject will be given a standardized pain medication prescription at their initial visit, and will be asked to keep track of how much pain medication they used each day, as well as to bring their pill bottle with them to the two-week follow-up appointment for a pill count. This information will be collected at the two-week follow-up appointment.
Time Frame: at 2 weeks
Population: Data is not available
Arm/Group | Silodosin | Tamsulosin
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Outpatient Treatment Failure
Description: Subjects will be given instructions at the initial visit to return to the emergency department immediately for signs and symptoms of infection or MET failure (fever, worsening pain, vomiting, lethargy, unsteadiness, syncope or inability to tolerate oral pain medications). These subjects will be considered to have failed outpatient treatment and will be removed from the study.
  Subjects who do not experience these issues but who still report having symptoms at the two-week follow-up visit will also be considered to have failed outpatient treatment.
Time Frame: at 2 weeks
Population: Data is not available
Arm/Group | Silodosin | Tamsulosin
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Adverse Hemodynamic Reaction
Description: Both tamsulosin and silodosin carry the possibility of causing orthostatic hypotension, which can manifest as unsteadiness, syncope, headache, and/or dizziness, especially when changing position from sitting/laying to standing. Subjects will be asked to assess themselves for these symptoms continuously from the initial visit, with serious reactions resulting in cessation of study medication. For reactions which are not serious, the information will be collected at the one-week follow-up call as well as the two-week follow-up visit.
Time Frame: at 2 weeks
Population: Data is not available
Arm/Group | Silodosin | Tamsulosin
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 0
Description: Data is not available: PI no longer at institution; attempts to contact unsuccessful
Arm/Group | Silodosin | Tamsulosin
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
0 Participants analyzed. PI has left the institution. Efforts made to contact the PI were unsuccessful. No study data available

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes